CLINICAL TRIAL: NCT04331691
Title: SPironolactone Versus Amiloride for Treatment of REsistant Hypertension (SPARE Trial): A Comparison of Home Blood Pressure
Brief Title: Comparison of Spironolactone and Amiloride on Home Blood Pressure in Resistant Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2019-1334
Record Dates: First submitted 2020-03-31; First posted 2020-04-02 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Resistant Hypertension
Keywords: Resistant Hypertension; Spironolactone; Amiloride; Home Blood Pressure Monitoring
MeSH Terms: interventions — Spironolactone; Amiloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spironolactone (Active Comparator): After randomization, this group will receive 12.5 mg of spironolactone daily. Subjects who did not reach the target blood pressure after 4 weeks of treatment should be increased to 25 mg of spironolactone. After 12 weeks of treatment, study will be end.
  Interventions: Drug: Spironolactone
- Amiloride (Experimental): After randomization, this group will receive 5 mg of amiloride daily. Subjects who did not reach the target blood pressure after 4 weeks of treatment should be increased to 10 mg of amiloride. After 12 weeks of treatment, study will be end.
  Interventions: Drug: Amiloride

INTERVENTIONS:
Drug: Spironolactone — After randomization, this group will receive 12.5 mg of spironolactone daily. Subjects who did not reach the target blood pressure after 4 weeks of treatment should be increased to 25 mg of spironolactone. After 12 weeks of treatment, study will be end.
  Arms: Spironolactone
Drug: Amiloride — After randomization, this group will receive 5 mg of amiloride daily. Subjects who did not reach the target blood pressure after 4 weeks of treatment should be increased to 10 mg of amiloride. After 12 weeks of treatment, study will be end.
  Arms: Amiloride

SUMMARY:
Resistant hypertension is defined as blood pressure that remains above goal despite concurrent use of three antihypertensive agents of different classes including diuretics. Patients with resistant hypertension has at least 1.5-fold higher cardiovascular risk than those with non-resistant hypertension. Therefore, controlling blood pressure is crucial in patients with resistant hypertension.

It has been unclear which antihypertensive agent should be added in patients who cannot reach target blood pressure despite use of three antihypertensive agents. There have been three randomized clinical trials that proved the efficacy of spironolactone in resistant hypertension, but they were small sized, comparison study to placebo. Recently published PATHWAY-2 study which compared the efficacy of spironolactone with placebo, doxazosin, and bisoprolol showed superiority of spironolactone in blood pressure lowering in patients with resistant hypertension. Thus, revised ACC/AHA and ESC/ESH guideline for arterial hypertension recommended spironolactone as the fourth agent for resistant hypertension. However, in real world, adherence to spironolactone may not be adequate because of adverse effect such as gynecomastia, hyperkalemia, and so on.

Recently, sub-study of PATHWAY-2 revealed that amiloride changes systolic blood pressure by -22.2 mmHg (95% CI, -24.7 to -19.7) which is comparable with the effect of spironolactone (-21.8 mmHg; 95% CI, -24.2 to -19.3). However, it was not randomized clinical trial to compare the effect between spironolactone and amiloride in patients with resistant hypertension.

This study aims to compare the effect of spironolactone and amiloride on home blood pressure in resistant hypertensive patients and to compare the rate of target blood pressure achievement between spironolactone and amiloride in resistant hypertensive patients.

DETAILED DESCRIPTION:
The subjects with office SBP of 130-180 mmHg with 3 antihypertensive medications of different classes including thiazide or thiazide-like diuretics and daytime average daytime SBP of ≥ 130 mmHg are enrolled in the 4-week run-in period. During run-in period, subjects will receive sevikar HCT (5/20/12.5 mg, 5/40/12.5 mg or 10/40/12.5 mg). After a 4-week run-in period, subjects who have uncontrolled average home SBP, defined as average SBP of ≥ 130 mmHg, will be randomized to either spironolactone or amiloride. 118 subjects will be randomly assigned to one of the two treatment groups. Subjects randomly assigned to one of the two treatment groups will receive 12.5 mg of spironolactone and the other group will receive 5 mg of amiloride. Subjects who did not reach the target blood pressure after 4 weeks of treatment should be increased to 25 mg of spironolactone or 10 mg of amiloride. After 12 weeks of treatment, study will be end.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-75
* Patients with resistant hypertension

  1. 1st screening: ven while taking three or more types of antihypertensive medications including diuretics without changing the dose for 1 month, the average office systolic blood pressure measured in three times is 130-180 mmHg and daytime systolic blood pressure is ≥130 mmHg.
  2. 2nd screening: An average systolic blood pressure of home blood pressure monitoring is ≥130 mmHg during the run-in period of antihypertensive drugs including diuretics (Sevikar HCT 5/20/12.5 mg, 5/40/12.5 mg or 10/40/12.5 mg).
* Patients with resistant hypertension who have agreed to participate in the study: when they have the ability to write a written consent in accordance with the Korean Good Clinical Practice (KGCP) and local laws.
* Patients who can change the currently used antihypertensive treatment to Sevikar HCT 5/20/12.5 mg, 5/40/12.5 mg or 10/40/12.5 mg without giving unacceptable risk (investigator's judgment)

Exclusion Criteria:

* White-coat uncontrolled hypertension
* Severe hypertension (WHO classification criteria grade 3 average diastolic blood pressure ≥ 110 mmHg or average systolic blood pressure ≥ 180 mmHg)
* Known cardiovascular disease (including stroke and TIA), including a history of angina, heart failure, myocardial infarction or revascularization, or cerebrovascular disease prior to 6 months
* Congestive heart failure of III-IV according to NYHA functional classification
* Clinically meaningful ventricular tachycardia, atrial fibrillation, atrial flutter, or other arrhythmia that the investigator has deemed clinically meaningful.
* Hypertrophic obstructive cardiomyopathy, severe obstructive coronary artery disease, aortic stenosis, hemodynamically significant aortic valve or stenosis on the mitral valve
* Renal insufficiency (basal estimated glomerular filtration rate (eGFR) <50 ml / min / 1.73m2)
* Hyperkalemia (> 5.0 mmol / L, which can be reconfirmed if errors are suspected in the results)
* Gastrointestinal diseases that can cause potential malabsorption the gastro-intestinal tract is severely narrowed; Kock pouch (a continent pouch formed by the terminal ileum after colectomy)
* Bile stasis or biliary obstruction
* liver disease or aspartate aminotransferase (AST) / alanine aminotransferase (ALT) levels > 2-fold the normal upper limit (ULN)
* Pregnant or fertile women who are not contraceptive or woman who are lactating
* Intolerant to test drug/drug group or its components
* Subjects who are currently participating in other clinical trials and who have taken other investigational product within the past month.
* Subjects who have condition or a disease that may impede the completion of the test, according to the investigator's opinion
* If assigned to treatment for this trial in the past
* Uncorrected sodium or fluid depletion
* History of drug or alcohol dependence within 6 months
* The combination of medications known to affect blood pressure, except those permitted by the protocol.
* Other clinical conditions that, as determined by the investigator, cannot be safely completed according to the protocol or that the investigational product cannot be safely used a history of secondary hypertension that cannot be corrected
* Taking spironolactone or amiloride within 4 weeks from the time of screening
* If discontinued due to side effects of spironolactone or amiloride

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
The difference between spironolactone versus amiloride for changes in home SBP from baseline to week 12. | week 12
  Comparison of the change of average home systolic blood pressure at week 12 from the introduction phase between spironolactone group and amiloride group

SECONDARY OUTCOMES:
target blood pressure achievement rates | week 12
  Comparison of achievement rate for target home and office BP between spironolactone group and amiloride group

CONTACTS AND LOCATIONS:
Overall Officials: Sungha Park, Principal Investigator — Severance Hospital
Locations (1):
- Severance Cardiovascular Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee CJ, Ihm SH, Shin DH, Jeong JO, Kim JH, Chun KH, Ryu J, Lee HY, Choi S, Lee EM, Choi JH, Kim KI, Shin J, Pyun WB, Kim DH, Park S, Williams B. Spironolactone vs Amiloride for Resistant Hypertension: A Randomized Clinical Trial. JAMA. 2025 Jun 17;333(23):2073-2082. doi: 10.1001/jama.2025.5129. PMID 40366680